CLINICAL TRIAL: NCT02577224
Title: A Randomised Controlled Trial to Explore the Effectiveness and Cost-effectiveness of a Patient-initiated Botulinum Toxin Treatment Model for Blepharospasm and Hemifacial Spasm Compared to Treatment as Usual
Brief Title: An RCT of a Patient-initiated Treatment Service for BEB and HFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Merz Pharmaceuticals (Industry); City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EZRD1024
Record Dates: First submitted 2015-05-08; First posted 2015-10-16 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Blepharospasm; Hemi Facial Spasm
Keywords: Patient-led care; Botulinum toxin; Dystonia; Randomised controlled trial; Acceptability
MeSH Terms: conditions — Blepharospasm; Dystonia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Participants randomized to the intervention group (patient-initiated treatment) will be asked to initiate their own treatment during the nine months they are taking part in the trial. Intervention group participants will receive information about when and how to initiate an appointment. Contact details for the service will be provided along with information on how quickly an appointment will be made, with whom and the procedure in the case of an emergency. All patients requesting an appointment will be booked in to the next available slot within the twice weekly ring-fenced nurse-led clinics. Any subsequent scheduled appointments will be cancelled and all future treatment will be initiated by the patient.
  Interventions: Other: Patient-initiated treatment
- Control (No Intervention): Participants in the control group will receive treatment as usual. This consists of scheduled appointments in the hospital-based nurse-led botulinum toxin clinic. The frequency with which these appointments takes place are based on clinical judgement, but tend to range between every 6 weeks to every 4 months.

INTERVENTIONS:
Other: Patient-initiated treatment — Please see Intervention Arm
  Arms: Intervention

SUMMARY:
Blepharospasm and hemifacial spasm are debilitating conditions which significantly impact on patient quality of life. Cyclical treatment with botulinum toxin injections offers temporary relief but the duration of treatment efficacy is variable. The standard model of patient care defines routine fixed- time based scheduled treatment cycles which may lead to unnecessarily frequent treatment for some patients and experience of distressing symptoms in others if symptoms return before the scheduled follow up period. The present study aims to compare a patient-initiated model of care, where patients determine treatment timing, with the standard model of care by using a two-arm randomised controlled trial design. It is expected that patients able to initiate their own treatment will experience less variation in disease severity and disability over a treatment cycle as they will be empowered to take the initiative when they feel they need to have treatment. A range of other outcomes will be assessed including: confidence and satisfaction in the service, depression, anxiety, quality of life and, illness and treatment beliefs. If the patient-led care model is shown to be effective in preventing distress and reducing disability in these populations; and is found to be acceptable to service users, this will have significant implications for service organisation across the NHS.

DETAILED DESCRIPTION:
Blepharospasm is a dystonia described by sustained, forced, involuntary closure of both eyelids, caused by muscle contraction. Hemifacial spasm occurs on one side of the face and can result in complete closure of one eye, and spasms across the cheek, face and neck. Hemifacial spasm, as its name implies, is unilateral, whereas blepharospasm always affects both eyes. Blepharospasm and hemifacial spasm are debilitating conditions, which carry the risk of functional blindness and can lead to appearance concerns, social embarrassment and isolation, depression and poor quality of life.[1-3]

Botulinum toxin is the treatment used in standard care to stop spasms, but results in a fluctuating pattern of relief and aggravation[4] and hence patients return for repeated injections. A recent systematic review indicated that the patient reported benefits of botulinum toxin in blepharospasm ranged from no improvement to 96% of patients reporting a significant relief in symptoms.[5] Evidence for the duration of benefit provided by repeated treatment is was also markedly inconsistant.[5] Although the definition of benefit did differ between studies in this review, research cannot explain such inconsistencies. Despite this a standardised treatment regimen, of injections on average 3 times a year, is currently used across all patients at Moorfields Eye Hospital and is typical throughout the UK. This may mean that some people are left experiencing debilitating symptoms until their next scheduled appointment and some are being seen too often, hence alternative models of care need to be considered.

Patient-centred care is at the forefront of the NHS,[6;7] reflecting the shift away from the paternalistic model of healthcare. Patients are now encouraged to take a more active role in knowing and managing their health, and this is especially important in conditions such as dystonia where the reality of living with the condition is demanding. As a result patient-led healthcare services are becoming increasingly more common and have the potential to address the inconsistencies found in the current botulinum toxin treatment regimen.

Research studies trialling patient-initiated services, where the patient rather than healthcare professional initiates treatment and care, have shown promise. These services provide patients with information on when and how to access services, rather than having regular scheduled appointments. A systematic review conducted by Whear et al[8] synthesised the evidence for this model of care across three conditions: irritable bowel disease, breast cancer and rheumatoid arthritis. Overall, there were few differences in psychological or health-related quality of life between those initiating their own outpatient follow-up appointments compared to standard care, despite in many cases patients having less contact with healthcare professionals. Patient and clinician satisfaction were also significantly greater in the patient-initiated services compared to regular appointment scheduling. Since this systematic review members of the research team have led on the development and evaluation of a patient-initiated follow-up service for patients with arthritis. Using a mixed methods study design the service was found to reduce healthcare utilisation in a RCT, without compromising clinical or psychosocial well-being, and was found to be acceptable to patients in the embedded qualitative study.[9]

Adopting a patient-led model of care could reduce discomfort and disability in patients with a short-term response to botulinum toxin and reduce unnecessary hospital visits and treatment for patients with a longer-term response. There is currently one patient-initiated, nurse-led botulinum toxin clinic running in the UK for patients with blepharospasm or hemifacial spasm,[10] but is yet to be evaluated in comparison to usual care. Due to the variable nature of treatment response blepharospasm and hemifacial spasm are appropriate conditions in which to evaluate a service of this nature. This study therefore, provides a unique opportunity to empower patients with dystonia to take control of their treatment and optimise the effects of botulinum toxin, by allowing them to seek treatment when they feel it is necessary rather than it being dictated by the clinical team, within the context of a methodologically robust evaluative.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemifacial spasm or blepharospasm
* Attending a hospital-based botulinum toxin clinic at Moorfields Eye Hospital NHS Foundation Trust.
* Patients stable on botulinum toxin treatment, defined as receiving toxin treatment at stable doses over two previous cycles and free from and side effects.
* Aged 18 years old and over.
* Capacity to give informed consent to participate in the study, judged by the Research Nurse.

Exclusion Criteria:

* Participants with significant co-morbidities (i.e. their predominant treatment is for another illness).
* Inability to communicate fluently in written and/or spoken English, to complete study measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Disease severity | 18 months
  For patients with blepharospasm and hemifacial spasm, disease severity and frequency of symptoms will be assessed using the Jankovic Rating Scale (JRS), a clinician completed measure. The JRS consists of two subscales that measure severity and frequency separately. A 2-point improvement in the JRS sum score is considered a clinically relevant improvement. For patients with hemifacial spasm an additional rating scale for severity and frequency of cheek involvement will be included, which has been recommended by the questionnaire developers.
Disability | 18 months
  The Blepharospasm Disability Index (BSDI)© is a patient self-report measure which asks patients' about six daily activities: reading, driving a vehicle, watching TV, shopping, walking and doing everyday activities. The measure is also recommended for use when assessing the impact of Botulinum toxin in hemifacial spasm. The measure has been found to possess good convergent validity with the JRS, good internal consistency (Cronbach's alpha = 0.88) and adequate test-retest reliability by its developers.
Patient satisfaction | 18 months
  Patient satisfaction will be measured using the 8-item Client Satisfaction Questionnaire (CSQ). The scale has good internal reliability, with Cronbach's alpha ranging from 0.93 to 0.93 and good construct validity

SECONDARY OUTCOMES:
Side effects | 18 months
  Individual side effects including ptosis, tearing, blurred vision, double vision, hematoma, foreign body sensation, will be recorded at each clinic visit. The total number of side effects will be recorded for each patient.
Confidence in system of care | 18 months
  Confidence in the system of care will be assessed using a 10cm visual analogue scale (VAS). Patients will be asked 'How confident are you that if you required treatment this system of care would be able to support you?' ranging from 'not at all confident' to 'completely confident'.
Patient quality of life | 18 months
  Quality of life will be measured using the Craniocervical dystonia questionnaire (CDQ-24) which was developed and validated in patients with blepharospasm, and has also been used with success in patients with hemifacial spasm. This 24 item measure assesses quality of life across five domains: stigma, emotional well-being, pain, activities of daily living and social/family life. The measure has been found to possess good internal consistency with Cronbach's alphas ranging from 0.77 to 0.89, good construct validity when compared who the SF-36, good discriminant validity and test retest reliability.
Mood | 18 months
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess mood. The HADS is a 14-item self-screening questionnaire for depression and anxiety in patients with physical health problems. The two 7-item subscales measure how a person has been feeling in the past week. The scale provides cut-off scores for the presence of potentially clinical levels of anxiety and depression. A systematic review of the HADS has confirmed the factor structure, found the cut-off points to be valid against clinical interviews, reports excellent internal consistency (Cronbach's alpha: anxiety 0.68-0.93; depression 0.67-0.90)
Illness perceptions | 18 months
  Illness perceptions are cognitive representations or beliefs that a patient has about their illness. These concepts will be measured using the revised illness perceptions questionnaire (IPQ-R), which has been widely used and is a valid and reliable measure.
Treatment beliefs | 18 months
  Beliefs about botulinum toxin will be measured using the Treatment Representations Inventory (TRI). A 27-item measure, consisting of four subscales including 'treatment-value', 'treatment-concerns', 'decision-satisfaction' and 'cure'.
Acceptability | 18 months
  Acceptability of the new patient-initiated service and standard care will be measured using the 7-item Acceptability Questionnaire developed by the study team.
Cost effectiveness | 18 months
  An adapted version of the Client Service Receipt Inventory (CSRI) has been employed, which has been widely employed in previous studies, particularly in the mental health setting. The impact of the service on direct and indirect costs will be estimated at the end of the trial period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ezra, MD FRCOph, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Kraft SP, Lang AE. Cranial dystonia, blepharospasm and hemifacial spasm: clinical features and treatment, including the use of botulinum toxin. CMAJ. 1988 Nov 1;139(9):837-44. PMID 3052771
- [Background] Muller J, Kemmler G, Wissel J, Schneider A, Voller B, Grossmann J, Diez J, Homann N, Wenning GK, Schnider P, Poewe W; Austrian Botulinum Toxin and Dystonia Study Group. The impact of blepharospasm and cervical dystonia on health-related quality of life and depression. J Neurol. 2002 Jul;249(7):842-6. doi: 10.1007/s00415-002-0733-1. PMID 12140667
- [Background] Reimer J, Gilg K, Karow A, Esser J, Franke GH. Health-related quality of life in blepharospasm or hemifacial spasm. Acta Neurol Scand. 2005 Jan;111(1):64-70. doi: 10.1111/j.1600-0404.2004.00357.x. PMID 15595940
- [Background] Jinnah HA, Berardelli A, Comella C, Defazio G, Delong MR, Factor S, Galpern WR, Hallett M, Ludlow CL, Perlmutter JS, Rosen AR; Dystonia Coalition Investigators. The focal dystonias: current views and challenges for future research. Mov Disord. 2013 Jun 15;28(7):926-43. doi: 10.1002/mds.25567. PMID 23893450
- [Background] Colosimo C, Tiple D, Berardelli A. Efficacy and safety of long-term botulinum toxin treatment in craniocervical dystonia: a systematic review. Neurotox Res. 2012 Nov;22(4):265-73. doi: 10.1007/s12640-012-9314-y. Epub 2012 Feb 23. PMID 22359151
- [Background] Whear R, Abdul-Rahman AK, Thompson-Coon J, Boddy K, Perry MG, Stein K. Patient initiated clinics for patients with chronic or recurrent conditions managed in secondary care: a systematic review of patient reported outcomes and patient and clinician satisfaction. BMC Health Serv Res. 2013 Dec 1;13:501. doi: 10.1186/1472-6963-13-501. PMID 24289832
- [Background] McBain H, Shipley M, Olaleye A, Moore S, Newman S. A patient-initiated DMARD self-monitoring service for people with rheumatoid or psoriatic arthritis on methotrexate: a randomised controlled trial. Ann Rheum Dis. 2016 Jul;75(7):1343-9. doi: 10.1136/annrheumdis-2015-207768. Epub 2015 Aug 19. PMID 26290587
- [Derived] Lawes-Wickwar S, McBain H, Brini S, Hirani SP, Hurt CS, Flood C, Dunlop N, Solly D, Crampton B, Newman SP, Ezra DG. A patient-initiated treatment model for blepharospasm and hemifacial spasm: a randomized controlled trial. BMC Neurol. 2022 Mar 17;22(1):99. doi: 10.1186/s12883-022-02603-7. PMID 35300599